CLINICAL TRIAL: NCT03417193
Title: Opioid Free Anesthesia in Major Spine Surgery: a Prospective, Double-blinded, Randomized, Controlled Trial
Brief Title: Opioid Free Anesthesia and Major Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lebanese American University (Other)
Responsible Party: Principal Investigator, Hanane Barakat, MD, Lebanese American University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LAUMCRH.HB1.11/Jan/2018
Record Dates: First submitted 2018-01-16; First posted 2018-01-31 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Opioid Use; Postoperative Pain; Spine Disease
Keywords: Lidocaine; Dexmedetomidine; Opioid-free
MeSH Terms: conditions — Pain, Postoperative; Spinal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioid based Anesthesia (Active Comparator): General anesthesia will be induced using Propofol , fentanyl , and Rocuronium . Ketamine will be administered on induction of anesthesia with the same dose to be repeated every hour. Anesthesia will be maintained with Remi-fentanyl , sevoflurane and nitrous oxide.
  Interventions: Drug: opioid free Anesthesia vs Opioid based Anesthesia
- Opioid Free Anesthesia (Active Comparator): -General anesthesia will be induced using dexmedetomidine and lidocaine started 10 minutes before induction, Propofol and Rocuronium . Ketamine will be administered on induction of anesthesia with the same dose to be repeated every hour. Anesthesia will be maintained with IV infusion of dexmedetomidine , lidocaine , sevoflurane and nitrous oxide.
  Interventions: Drug: opioid free Anesthesia vs Opioid based Anesthesia

INTERVENTIONS:
Drug: opioid free Anesthesia vs Opioid based Anesthesia — Compare the opioid based anesthesia with Fentanyl and Remifentanyl to opioid free anesthesia with dexmedetomidine and lidocaine and their effect on postoperative pain.

SUMMARY:
This study compares the intraoperative opioid free anesthesia approach in multilevel spine posterior instrumentation surgery to a conventional opioid-based anesthesia. Half of participants will receive opioid free anesthesia with dexmedetomidine, lidocaine and ketamine while the other half will receive opioid based anesthesia with fentanyl, remi-fentanyl and ketamine

DETAILED DESCRIPTION:
Opioid analgesics are commonly used in clinical practice for per and postoperative pain treatment. However their use is associated with a lot of undesirable effects. From this comes the idea of using opioid free anesthesia intra-operatively in an attempt to decrease opioids postoperative use and accordingly, their associated side effects.

Intravenous (IV) lidocaine has been found to have analgesic, antihyperalgesic, and anti-inflammatory properties. It was found to significantly improve postoperative pain, when its intraoperative use was compared with placebo .

Dexmedetomidine is a selective alpha-two adrenergic receptor agonist that has antinociceptive, analgesic, opioid sparing and sedative properties. Similar to lidocaine, dexmedetomidine was shown to lower postoperative pain, opioid consumption and accordingly, opioid related side effects.

ELIGIBILITY:
Inclusion Criteria:

* Age group: 18-80 years old
* American Society of Anesthesiologists (ASA )class I, II and III
* Elective spine posterior instrumentation surgery of at least two levels.

Exclusion Criteria:

* Renal, hepatic or cardiac insufficiency.
* Alcohol or drug abuse.
* Psychiatric disease.
* Allergy or contraindication to any of the study drugs.
* Inability to comprehend pain assessment or inability to use a Patient Controlled Analgesia (PCA) device.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2023-02-16 (Actual); Study Completion 2023-02-16 (Actual)

PRIMARY OUTCOMES:
Postoperative morphine consumption | 48 hours
  After the surgery the patient will go to the PACU (Post Anesthesia Care Unit). the patient will receive morphine if the pain score is more than 4. the total dose of morphine in mg (milligrams) will be documented. Before discharge from the PACU, the patient will have a PCA (Patient Controlled Analgesia) morphine,All attempts and given values of morphine In mg obtained from the PCA machine will be documented at 0, 1, 2, 4, 6, 12, 18, and 24 hours and every 6 hours thereafter up to 48 hours post surgery..
  And the total amount of morphine in mg will be calculated for 48 hours

SECONDARY OUTCOMES:
Postoperative morphine Side effects: Sedation score . | 48 hours post operative.
  -Sedation score: 0 alert
  1. Mild, drowsy , easy to awake
  2. moderate, easy to arouse
  3. Severe: somnolent difficult to arouse 4:sleeping The Sedation score will be documented at 0, 1, 2, 4, 6, 12, 18, and 24 hours and every 6 hours thereafter up to 48 hours.
Postoperative morphine Side effects:Respiratory depression | 48 hours
  Assess the respiratory rate : The number of breaths per minute. In practice, the respiratory rate is usually determined by counting the number of times the chest rises or falls per minute.
  The respiratory rate will be documented at 0, 1, 2, 4, 6, 12, 18, and 24 hours and every 6 hours thereafter up to 48 hours.
Postoperative morphine Side effects: Nausea vomiting | 48 hours
  Degree of nausea vomiting using the verbal rating score from 0 to 10 : 0= no nausea/ Vomiting, 10: worst possible nausea vomiting.
  The degree of nausea vomiting will be documented at 0, 1, 2, 4, 6, 12, 18, and 24 hours and every 6 hours thereafter up to 48 hours.
Postoperative morphine Side effects: Itching | 48 hours
  Itching: presence or absence The presence or absence of itching will be documented at 0, 1, 2, 4, 6, 12, 18, and 24 hours and every 6 hours thereafter up to 48 hours.
Postoperative pain score | 48 hours post operative.
  Measure the pain score using the Visual Analogue Scale (VAS), The Visual Analogue Scale (VAS) consists of a straight line with the endpoints defining extreme limits such as 'no pain at all' and 'pain as bad as it could be' The patient is asked to mark his pain level on the line between the two endpoints. The distance between 'no pain at all' and the mark then defines the subject's pain. The score ranges from 0 to 100 mm. A higher score indicates greater pain intensity. The distribution pain is the following:no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm).Postoperative pain will be measured using Verbal Analogue Scale (VAS) at 0, 1, 2, 4, 6, 12, 18, and 24 hours to be repeated every 6 hours thereafter up to 48 hours post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hanane MD, Principal Investigator — Lebanese American University/ LAU Medical Center
Locations (1):
- LAU Medical Center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No